CLINICAL TRIAL: NCT04697004
Title: A Randomized, Multi-Center, Prospective, Safety and Efficacy Study Comparing the Outcome of Total Reverse Shoulder Arthroplasty (RSA) with SMR Stemless Reverse Vs SMR Reverse Shoulder System
Brief Title: SMR Stemless Reverse Vs SMR Reverse Shoulder System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Limacorporate S.p.a (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-34
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2023-10

CONDITIONS: Arthroplasty, Replacement
Keywords: Shoulder Joint; Shoulder Replacement; Arthritis with rotator cuff tear; Post traumatic fracture sequele; Severe osteoarthritis and rotator cuff deficiency; Significant glenoid or socket side bone deformed or loss; Reoccurrence of instability or chronic shoulder dislocation; Severe osteoarthritis and stiff shoulder
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: The 200 randomized subjects will be randomized 1:1 to SMR Stemless Reverse and SMR Reverse Shoulder System.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- SMR Stemless Reverse (Experimental)
  Interventions: Device: Investigational Arm: SMR Stemless Reverse
- SMR Reverse Shoulder System (Active Comparator)
  Interventions: Device: Control Arm: SMR Reverse Shoulder System

INTERVENTIONS:
Device: Investigational Arm: SMR Stemless Reverse — The SMR Stemless Reverse is intended for total, primary shoulder joint replacement by reducing pain and restoring shoulder articular mobility function.
  Arms: SMR Stemless Reverse
Device: Control Arm: SMR Reverse Shoulder System — Conventional stemmed shoulder prostheses are commonly used in the clinical practice.
  Arms: SMR Reverse Shoulder System

SUMMARY:
The SMR Stemless Reverse is intended for total, primary shoulder joint replacement by reducing pain and restoring shoulder articular mobility function. This is a prospective, multi-center, randomized, controlled trial to demonstrate non-inferiority of the SMR Stemless Reverse to the SMR Reverse Shoulder System.

Patients with joint dysfunction who continue to experience significant symptoms despite an appropriate course of non-operative management are eligible. Patients will be considered enrolled into the study when an ICF has been signed, all inclusion criteria are met and no exclusion criteria are present including intraoperative exclusion criteria, and the patient is randomized into either the SMR Stemless Reverse (investigational) group, the SMR Reverse Shoulder System (control) group or is part of the roll-in population. Enrollment is expected to take approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22 years of age
2. Skeletally mature as evident by scapula and proximal humerus closure
3. Candidate for primary total shoulder replacement in a grossly rotator cuff deficient joint with severe arthropathy (disabled shoulder), when clinical indications based on physical exam and medical history including one or more of the following:

   1. Arthritis with rotator cuff tear not reparable
   2. Irreparable rotator cuff tear
   3. Rotator cuff tear arthropathy
   4. Severe osteoarthritis and rotator cuff deficiency or stiff shoulder
   5. Significant glenoid or socket side bone deformed or loss
   6. Reoccurrence of instability or a chronic shoulder dislocation
   7. Any other medical reason that the investigator determine that subject is a good candidate for a reverse total shoulder arthroplasty

Exclusion Criteria:

1. BMI > 40 kg/m2
2. Previous contralateral shoulder surgery within 3 months of enrollment or that requires active treatment (i.e. surgery or brace)
3. Had surgery in the targeted shoulder within last 12 months of enrollment, except diagnostic arthroscopy without procedures
4. Had surgery in lower limbs (such as hip or knee) within last 6 months of enrollment
5. Corticosteroid injections in the ipsilateral shoulder within 3 months of enrollment
6. Complete deltoid muscle insufficiency
7. Glenoid retroversion great than 25 degrees based off a 2D axial CT scan
8. History of/or signs and/or symptoms of local or systemic infection including but not limited to septicemia; osteomyelitis
9. Neurologically confirmed nerve lesion compromising shoulder joint function
10. Poor meta-epiphyseal bone stock compromising stability of the implant including but not limited to humeral head fracture, iatrogenic glenoid fracture, severe osteoporosis
11. Metabolic disorders which may impair fixation and stability of the implant including but not limited to uncontrolled diabetes mellitus with an HbA1C > 7.5%
12. Extended bone loss after previous surgery defined as: complete bone loss of greater and lesser tuberosity
13. Meta-epiphyseal bony defect (including large cyst)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint-Constant Murley Score | 24 Months
  The primary efficacy endpoint is to assess successful clinical outcomes by Constant-Murley Score (CMS) adjusted for gender and age at month 24 defined as an increase in CMS of at least 15 points over baseline CMS.
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The higher the score, the higher the quality of the function.
Primary Safety Endpoint-Absence of revisions, reoperations, and implant loosening. | 24 Months
  * Revisions - A revision is a procedure that adjusts, modifies, or removes part of the original implant configuration, with or without replacement of a component. This may include removing a component of a joint implant.
  * Reoperations - A reoperation is any surgical procedure involving the repaired shoulder that does not include removal, modification, or addition of any components to the investigational device (e.g., drainage of a hematoma at the surgical site).
  Radiographic: Implant Loosening
  * A humeral component is considered to be at risk for loosening when a radiolucent line >2 mm is present in four (4) or more of the eight (8) zones or if there is conclusive evidence of migration or tilt of the component.
  * A glenoid component is considered to be at risk for loosening in case of conclusive evidence of a migration or tilt of the component or in presence of a circumferential radiolucent line of at least 2 mm around the glenoid component.

SECONDARY OUTCOMES:
Secondary Efficacy Measure-Constant-Murley Score | 3, 6, and 12 month visits
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The higher the score, the higher the quality of the function.
Secondary Efficacy Measure-American Shoulder and Elbow Surgeons Shoulder Score (ASES) | 3, 6, 12 and 24 month visits
  The ASES questionnaire is composed of both a physician-rated component and a patient-reported component. The patient questions focus on joint pain, instability, and activities of daily living. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Secondary Efficacy Measure-Simple Shoulder Test (SST) | 3, 6, 12 and 24 month visits
  Simple Shoulder Test (SST) is a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. The answers to these questions provides a standardized way of recording the function of a shoulder before and after treatment. The difference between the shoulder function before treatment and after the recovery period is the effectiveness of the treatment.
Secondary Efficacy Measure-EQ-5D-5L | 3, 6, 12 and 24 month visits
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. This tool also has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable condition of health.
Secondary Efficacy Measure-Range of Motion (ROM) | 3, 6, 12 and 24 month visits
  will be summarized using the mean, standard deviation, sample size, median and minimum and maximum scores and will be presented separately for the SMR Stemless Reverse and SMR Reverse Shoulder System implant groups.
Secondary Efficacy Measure-Single Assessment Numeric Evaluation (SANE) | 3, 6, 12 and 24 month visits
  The Single Assessment Numeric Evaluation (SANE) is a simple, one-question patient-reported outcome measures. Patient reported outcome measures (PROMs) quantify symptoms and limitations in people with musculoskeletal illness. The Single Assessment Numeric Evaluation (SANE) is a patient rating from 0-100. Patients rate their current illness score in relation to their pre-injury baseline.
Secondary Safety Measure-Serious Procedure or Device Related Adverse Events | From enrollment to the final study visit (24 months)
  Serious Procedure or Device Related Adverse Events, device deficiencies, malfunctions and use errors at all follow-up time points
Secondary Safety Measure-Absence of Subsequent Secondary Surgical Interventions | From enrollment to the final study visit (24 months)
  Absence of:
  * Removals - A removal is a procedure where all of the original system configuration is removed with or without replacement due to, for example, mechanical failure of the device, pain, or infection.
  * Supplemental Fixations - A supplemental fixation is a procedure in which additional instrumentation not under study in the protocol is implanted (e.g., supplemental placement of a rod/screw)
Secondary Safety Measure-Radiographic: Standard CT and x-ray scans | From enrollment to the final study visit (24 months)
  Presence/absence of and fracture, radiolucent , migration, mal-alignment or loss of reduction or fixation.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Garrigues, M.D., Principal Investigator — Rush Orthopedics
Locations (11):
- United States (11):
  - Cedars-Sinai Kerlan-Jobe Institute, Los Angeles, California
  - Western Orthopaedics, Denver, Colorado
  - Levy Shoulder Center, Boca Raton, Florida
  - AdventHealth, Orlando, Florida
  - Rush Orthopaedics, Chicago, Illinois
  - Upstate Orthopedics, East Syracuse, New York
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rothman Orthopaedic, Philadelphia, Pennsylvania
  - Guthrie, Sayre, Pennsylvania
  - University of Texas- Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No